CLINICAL TRIAL: NCT06869226
Title: A Multicenter Phase II Clinical Study of Neoadjuvant Use of Camrelizumab in Combination With Chemotherapy for Organ Preservation in Esophageal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024YJZ151
Record Dates: First submitted 2025-03-05; First posted 2025-03-11 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-03

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — camrelizumab; 130-nm albumin-bound paclitaxel; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab+chemotherapy (Experimental)
  Interventions: Drug: Camrelizumab + Nab-paclitaxel + Cisplatin

INTERVENTIONS:
Drug: Camrelizumab + Nab-paclitaxel + Cisplatin — Three cycles of neoadjuvant therapy with camrelizumab (200 mg/dose D1, IV, Q3W)+Nab-paclitaxel(260 mg/m2 D1，IV，Q3W)+Cisplatin(75 mg/m2 D1，IV，Q3W); for patients with organ preservation intent entered into the watchful waiting strategy group and received radiotherapy (50.4 Gy/28 doses), with camrelizumab maintenance therapy for 4-12 weeks after the end of radiotherapy, and a total of up to one year of camrelizumab.

SUMMARY:
This is a multicenter phase II clinical study to explore the efficacy, safety, and organ preservation feasibility of camrelizumab in combination with chemotherapy for resectable esophageal squamous carcinoma in patients with histologically and pathologically confirmed resectable esophageal squamous carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily enrolled in this study, signed the informed consent form, had good compliance, and could cooperate with follow-up visits;
2. esophageal cancer diagnosed by histopathology; clinical staging of cT1b-cT2 N+ M0 or cT3, any N, M0 (according to AJCC 8th edition);
3. Age 18-75 years old, male or female;
4. ECOG PS 0-1;
5. measurable tumor lesions or non-measurable lesions that can be evaluated;
6. not having received any previous anti-tumor therapy for esophageal cancer, including radiotherapy, chemotherapy, surgery, etc;
7. Normal or mildly to moderately abnormal lung function (VC%>60%, FEV1>1.2L, FEV1%>40%, DLco>40%) that can tolerate esophageal cancer resection;
8. No contraindications to surgery;
9. function of vital organs meets the following requirements (excluding the use of any blood components and cell growth factors within 14 days): (1) Normal bone marrow reserve function with white blood cell (WBC) ≥3.0×109/L; neutrophil count (NEUT) ≥1.5×109/L, platelet count (PLT) ≥100×109/L, hemoglobin (Hb) ≥90g/L; (2) Normal renal function with serum creatinine (SCr) ≤1.5 times upper limit of normal (ULN) or creatinine clearance ≥60 ml/min (Cockcroft-Gault formula); (3) Normal liver function with total bilirubin (TBIL) ≤1.5 times the upper limit of normal (ULN); and an albumin transaminase (AST) or alanine transaminase (ALT) level ≤2.5 times the upper limit of normal (ULN); (4) Normal coagulation function with International Normalized Ratio (INR) ≤ 1.5 times the upper limit of normal (ULN) and Activated Partial Thromboplastin Time (APTT) ≤ 1.5 times the upper limit of normal (ULN).
10. Patients with potential childbearing potential are required to use a medically approved contraceptive method (e.g., IUD, birth control pills, or condoms) during and for 6 months after the end of the study treatment period; must have had a negative serum HCG or urine HCG test for 72 h prior to study entry; and must not be breastfeeding.

Exclusion Criteria:

1. Presence of locally advanced unresectable (regardless of stage) or metastatic disease (stage IV);
2. Exclude patients with cervical segment esophageal cancer;
3. Previous history of allergy to monoclonal antibodies, any component of karelizumab, albumin-bound paclitaxel, carboplatin or other platinum drugs;
4. patients with moderate or greater chest and back pain and risk of esophageal perforation.
5. have received or are receiving any of the following treatments in the past: (1) any radiotherapy, chemotherapy, or other antineoplastic agents directed against the tumor; (2) Treatment with immunosuppressive drugs, or systemic hormonal drugs for immunosuppression (doses >10 mg/day prednisone or equivalent) within 2 weeks prior to first use of study drug; inhaled or topical steroids and adrenocorticotropic hormone replacement at doses >10 mg/day prednisone or equivalent are permissible in the absence of active autoimmune disease; (3) Received a live attenuated vaccine within 4 weeks prior to first use of study drug; (4) Major surgery or severe trauma within 4 weeks prior to first use of study drug;
6. Have any active autoimmune disease or history of autoimmune disease, including but not limited to: interstitial pneumonitis, enteritis, hepatitis, pituitary gland inflammation, vasculitis, nephritis, hyperthyroidism, hypothyroidism (may be considered for inclusion after hormone replacement therapy); patients with psoriasis or childhood asthma/allergies that have been in complete remission and do not require any interventions in adulthood may be considered for inclusion, but patients requiring bronchial Patients who require medical intervention with bronchodilators may not be included;
7. a history of immunodeficiency, including a positive HIV test, or other acquired or congenital immunodeficiency disease, or a history of organ transplantation or allogeneic bone marrow transplantation;
8. the presence of clinically uncontrolled cardiac conditions or diseases, including but not limited to, such as (1) NYHA class II or higher heart failure, (2) unstable angina pectoris, (3) myocardial infarction within 1 year, and (4) clinically significant supraventricular or ventricular arrhythmia that is not clinically intervened with or remains poorly controlled after clinical intervention;
9. a serious infection (CTCAE grade 2) such as severe pneumonia requiring hospitalization, bacteremia, or infectious co-morbidities within 4 weeks prior to the first use of study drug; except for prophylactic antibiotic use if baseline chest imaging suggests the presence of active pulmonary inflammation, signs and symptoms of infection within 14 days prior to the first use of study drug, or the need for treatment with oral or intravenous antibiotics;
10. the presence of active tuberculosis infection by history or CT scan, or a history of active tuberculosis infection within 1 year prior to enrollment, or a history of active tuberculosis infection more than 1 year ago without regular treatment
11. Presence of active hepatitis B HBV DNA ≥ 2000 IU/mL or 104 copies/mL hepatitis C (hepatitis C antibody positive and HCV RNA above the lower detection limit of the analytical method);
12. other malignancies diagnosed within 5 years prior to first use of study drug, unless malignancies with a low risk of metastasis or risk of death (5-year survival > 90%), such as adequately treated basal cell carcinoma of the skin or squamous cell skin carcinoma or carcinoma of the cervix in situ, may be considered for enrollment
13. Pregnant or lactating females;
14. In the judgment of the investigator, there are other factors that may lead to forced termination of the study in the middle of the study, such as suffering from other serious illnesses (including psychiatric illnesses) that require comorbid treatment, alcoholism, drug abuse, family or social factors that may affect the safety of or compliance with the subject.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 283 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | about 2 years
  The length of time between signing the informed consent form and the occurrence of any of the following events: disease progression, disease recurrence, or death from any cause

SECONDARY OUTCOMES:
Clinical complete remission (cCR) rate | about 2 years
  Defined as the proportion of subjects who achieved CR as assessed according to RECIST 1.1 and whose endoscopic biopsies were free of residual tumor;
Pathologic complete remission (pCR) rate | about 2 years
  Defined as no residual tumor cells after evaluation of the resected tumor tissue and regional lymph.
Progression-free survival (PFS) in subjects with organ preservation strategies | about 2 years
  From the time of dosing until tumor recurrence, including local recurrence or distant metastasis or death from any cause, based on imaging evaluation or tissue biopsy evidence, whichever occurs first;
Overall survival (OS) in subjects with organ preservation strategies | about 2 years
  Time from administration to death from any cause
Adverse Events (AE) | about 2 years
  Incidence and grade (including serious adverse events and immunization-related adverse events), as determined by NCI-CTCAE 5.0 criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Cancer Hospital, Beijing, China